CLINICAL TRIAL: NCT00109278
Title: A Comparison of the Safety, Tolerability, and Immunogenicity of V205C Manufactured From the 2003 Measles Stock Seed With Recombinant Human Albumin (rHA) Versus Currently Licensed V205C Manufactured From the 1967 Measles Stock Seed With Human Serum Albumin (HSA) in Healthy Children 12 to 18 Months of Age
Brief Title: A Measles, Mumps, and Rubella Investigational Vaccine Trial (V205C-010)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V205C-010; 2005_016
Record Dates: First submitted 2005-04-26; First posted 2005-04-26 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Measles
Keywords: Prevention of Measles
MeSH Terms: conditions — Measles | interventions — Rubella Vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Biological: V205C, measles, mumps, and rubella virus vaccine live
Biological: Comparator: Measles, Mumps, and Rubella Virus Vaccine Live

SUMMARY:
The purpose of this study is to test the safety of a measles, mumps, and rubella study vaccine made from a new measles stock seed (a component of the vaccine made in 2003) with rHA (recombinant human albumin).

DETAILED DESCRIPTION:
The duration of treatment is 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children 12 to 18 months of age.

Exclusion Criteria:

* Previous receipt of measles, mumps, rubella and/or varicella vaccine.
* Prior infection or exposure to (within last 4 weeks) measles, mumps, rubella, varicella and/or zoster.
* Any medical condition that might interfere with the immune response to the given vaccines (including HIV infection and/or cancer) or has undergone immunosuppressive (weakens your body's ability to fight infection) therapy.
* History of seizures (convulsions)
* Allergies to any component of the vaccine, including sorbitol, gelatin, or neomycin.
* A recent (within the last 3 days) illness resulting in a fever (underarm temperature greater than 99.5° F [37.5° C]).

Ages: 12 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1100 (Actual)
Dates: Start 2004-10; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Antibody response rate to measles at 6 weeks postvaccination

SECONDARY OUTCOMES:
Geometric mean titers to measles by ELISA at 6 weeks postvaccination

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html